CLINICAL TRIAL: NCT07185503
Title: The Efficacy and Safety of Liposomal Amphotericin B 3-5mg/kg Combined With Posaconazole/Isavuconazole for the Treatment of Mucormycosis in Patients With Hematologic Malignancies
Brief Title: Liposomal Amphotericin B Plus Posaconazole/Isavuconazole for Mucormycosis in Hematologic Malignancies: Efficacy and Safety
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2025004
Record Dates: First submitted 2025-08-01; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mucormycosis in Hematologic Malignancies
Keywords: Mucormycosis; Hematologic Malignancies; Liposomal Amphotericin B; posaconazole or isavuconazole
MeSH Terms: conditions — Mucormycosis; Hematologic Neoplasms | interventions — liposomal amphotericin B; posaconazole; isavuconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single-arm,multi-center real-world study: This is a single-arm study where all participants receive the same treatment. Participants will be treated with a combination antifungal regimen comprising:
  1. Liposomal Amphotericin B (L-AmB):
     Dose: 3-5 mg/kg/day administered intravenously (IV). Duration: Daily infusions until clinical stability, with adjustments permitted based on disease severity and tolerability.
  2. Posaconazole or Isavuconazole:
  Formulations: Oral tablets or intravenous (IV) formulations. Dosing: Loading dose: As per product labeling. Maintenance dose: 300 mg (posaconazole) or 200 mg (isavuconazole) once daily. Duration: Continued orally after discontinuation of L-AmB, per clinical judgment.
  Interventions: Drug: liposomal amphotericin B (3-5 mg/kg/day) combined with posaconazole/isavuconazole

INTERVENTIONS:
Drug: liposomal amphotericin B (3-5 mg/kg/day) combined with posaconazole/isavuconazole — The intervention in this study is a tailored antifungal regimen combining liposomal amphotericin B (L-AmB) (3-5 mg/kg/day IV) with posaconazole or isavuconazole (300 mg/200 mg daily, oral or IV), designed to optimize efficacy and safety in immunocompromised adults with blood cancers and mucormycosis. Dosing and duration are personalized based on clinical response, immune recovery, and organ function, with a focus on transitioning to oral therapy to reduce hospitalization. The study emphasizes rigorous safety monitoring, prohibited unauthorized antifungal co-medications, and explores prognostic factors to advance treatment strategies for this high-risk population.

SUMMARY:
This clinical trial, a single-arm prospective study, aims to evaluate the efficacy and safety of liposomal amphotericin B (3-5 mg/kg/day) combined with posaconazole/isavuconazole in treating adult patients with malignant hematological diseases complicated by mucormycosis. The primary objectives are to determine the proportion of patients achieving complete or partial resolution of mucormycosis symptoms and to identify prognostic factors influencing survival outcomes. Participants will receive the combination therapy, undergo regular monitoring of symptoms, adverse events, and disease progression via radiological and laboratory assessments, and complete follow-up visits to track long-term survival. The study will analyze composite response rates, treatment-related adverse events, and survival data to refine therapeutic strategies for this high-risk population.

DETAILED DESCRIPTION:
This research aims to test whether combining two antifungal medications-liposomal amphotericin B (given through an IV) and either posaconazole or isavuconazole (available as IV or oral pills)-can effectively and safely treat adults with blood cancers (like leukemia or lymphoma) who develop a severe fungal infection called mucormycosis. Current guidelines often recommend amphotericin B-based therapies, but optimal dosing, combinations, and treatment duration remain unclear. This study will provide critical data on whether a regimen of liposomal amphotericin B (3-5 mg/kg/day) paired with newer antifungals (posaconazole/isavuconazole) can enhance outcomes. It will also identify which patient characteristics (e.g., age, cancer type, recovery speed) most strongly affect survival, helping doctors personalize care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a hematologic malignancy (e.g., leukemia, lymphoma, myelodysplastic syndrome).
* Proven, probable, or possible invasive mucormycosis according to the 2019 European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) criteria.
* Age ≥18 years and ≤65 years at enrollment.
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2.
* No clinically significant organ dysfunction (e.g., renal, hepatic, cardiac) at screening that would preclude protocol-defined therapies.
* Ability to understand the study procedures and provide voluntary written informed consent.

Exclusion Criteria:

* Prior treatment with non-liposomal amphotericin B formulations (e.g., amphotericin B deoxycholate) for ≥4 days.
* Documented hypersensitivity, severe immediate allergic reaction, or intolerance to liposomal amphotericin B.
* History of a second malignancy (other than the index hematologic malignancy) treated within the past 3 years.
* Active HIV infection, hepatitis B virus (HBV) infection (HBsAg-positive), hepatitis C virus (HCV) infection (RNA-positive), or syphilis.
* Psychiatric disorders, cognitive impairment, or other conditions impairing compliance with study procedures or assessments.
* Pregnant females, breastfeeding females, or individuals of reproductive potential unwilling to use effective contraception during treatment and for ≥3 months post-therapy.
* Serum creatinine ≥2.0 × upper limit of normal (ULN).
* Liver transaminases (ALT/AST) or alkaline phosphatase ≥5.0 × ULN.
* Total bilirubin ≥3.0 × ULN (isolated bilirubin ≥3.0 × ULN is permitted if due to Gilbert's syndrome or hemolysis).
* Patients deemed ineligible by the investigator due to medical, ethical, or logistical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mucormycosis in Hematologic Malignancies patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Composite Response Rate at End of liposomal amphotericin B (L-AmB) (3-5 mg/kg/day IV) Therapy | Assessed immediately after discontinuation of liposomal amphotericin B therapy.
  The proportion of participants achieving a composite response, defined as the complete or partial resolution of mucormycosis-related clinical symptoms, radiological improvement (e.g., reduction in lesion size on CT/MRI), and microbiological clearance (e.g., negative fungal cultures or biomarkers).

SECONDARY OUTCOMES:
Survival Rate at Key Time Points | Day 84
  Proportion of participants alive at (1) end of liposomal amphotericin B (L-AmB) therapy, (2) 42 days post-therapy, and (3) 84 days post-therapy. Survival is defined as being free from death due to any cause.
Time to Favorable Overall Response | From date of enrollment until the date of first documented response, assessed up to 84 dsys.
  Duration from study enrollment to achievement of a favorable overall response (complete or partial resolution of mucormycosis symptoms, radiological improvement, and microbiological clearance).
Length of Hospitalization | Measured immediately after the intervention
  Total number of days participants spend hospitalized from enrollment until discharge or death.
Safety and Tolerability Profile | Measured immediately after the intervention
  Incidence and severity of treatment-emergent adverse events (TEAEs), including nephrotoxicity, hepatotoxicity, infusion reactions, and electrolyte abnormalities, graded per CTCAE v5.0 criteria.

OTHER OUTCOMES:
Association Between Baseline/Treatment Features and Survival Outcomes | Data analyzed post-study completion, using baseline and longitudinal data collected throughout the trial (6-18 months post-enrollment).
  Exploratory analysis to evaluate correlations between pre-treatment (e.g., neutrophil count, cancer stage, comorbidities), intra-treatment (e.g., time to clinical stability, antifungal dose adjustments), and radiological features (e.g., lesion size, anatomical location) with overall survival and disease relapse. Statistical methods (e.g., Cox regression, machine learning) will identify potential prognostic biomarkers or clinical predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Sizhou Feng, Study Director — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (9):
- China (9):
  - The Second Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Tianjin First Central Hospital, Tianjin
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin
  - Second Hospital of Tianjin Medical University, Tianjin
  - Tianjin Haihe Hospital, Tianjin
  - Tianjin Union Medical Center of Nankai University, Tianjin

IPD SHARING:
Plan to Share IPD: No